CLINICAL TRIAL: NCT00302133
Title: Optimizing Pharmacotherapy for Bipolar Alcoholics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ihsan Salloum, Professor of Psychiatry, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RO1-AA015385-01 -Salloum; R01AA015385-01 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Bipolar Disorder; Alcohol Dependence
Keywords: Alcoholism Bipolar Disorder Pharmacotherapy Naltrexone
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone add on to valproate (Experimental): Naltrexone hydrochloride 50 mg capsule daily for 12 weeks add on to valproate
  Interventions: Drug: Naltrexone hydrochloride
- Placebo add on to valproate (Placebo Comparator): Placebo comparator one capsule daily for 12 weeks add on to valproate
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naltrexone hydrochloride — Naltrexone hydrochloride 50 mg capsule daily for 12 weeks
  Other Names: Revia
  Arms: Naltrexone add on to valproate
Other: Placebo — Placebo arm
  Arms: Placebo add on to valproate

SUMMARY:
The purpose of this study is to test the efficacy of naltrexone and valproate in the treatment of comorbid bipolar disorder and alcohol dependence.

DETAILED DESCRIPTION:
Bipolar disorder has the highest rate of association with alcohol and other substance use disorders. This complex clinical presentation is asociated with severe disabilities,morbidity and heightened risk for suicide. There is a significant gap in our knowledge regarding effective treatment interventions for this high risk clinical population. This proposal will test the efficacy of a promising pharmacological approach for the treatment of comorbid alcohol dependence and bipolar disorder. We propose a randomized, double blind, placebo controlled 12-week trial to test the efficacy of valproate plus naltrexone vs. valproate alone in decreasing alcohol use and stabilizing mood symptoms among patients with comorbid alcohol dependence and bipolar disorder. All participants receive supportive psychosocial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet Diagnostic and Statistical Manual-IV (DSM-IV) criteria for current alcohol dependence and a concurrent bipolar disorder

Exclusion Criteria:

* 1) Schizophrenia, schizoaffective and any nonbipolar psychotic disorder, unipolar major depression, primary anxiety disorder,mental retardation and signs of impaired cognitive functioning.
* 2) Opiate dependence, abuse, or on opioid maintenance treatment for any reason and those with positive urine screen for opiate.
* 3)Current DSM-IV criteria for dependence on substances other that alcohol, cannabis,nicotine or caffeine.
* 4) Neurological conditions including epilepsy, history of brain injury,encephalitis or any organic brain syndrome or documented focally abnormal EEG.
* 5)Medical conditions including severe cardiac, liver, kidney, endocrine, hematologic, or other impairing medical conditions, or impending surgery
* 6)Pregnancy
* 7)Inability or unwillingness to use contraceptive methods
* 8)Any medical condition or other reason that in the opinion of the investigator would prevent the subject from completing the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-05; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan M Salloum, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sample drawn from University-based mental health services, community treatment programs and advertisement
Pre-assignment Details: Total telephone screened included 696 inquiries: 517 excluded for not meeting initial screen criteria; 91 excluded for lost to follow-up with continuing screening; 88 enrolled into the study.
  Of the 88 enrolled, 35 excluded for not meeting the inclusion criteria; 35 were lost to follow-up before group assignment.
Groups:
- Naltrexone: Naltrexone add on to valproate open label
  Naltrexone Hydrochloride 50 mg daily for 12 weeks
- Placebo: Placebo add on to valproate open label
  Placebo one capsule daily for 12 weeks
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 9 | 9
Completed | 5 | 5
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Naltrexone: Naltrexone add on to valproate open label
  naltrexone add on to open label valproate: naltrexone 50 mg/day for 12 weeks add on to open label valproate
- Placebo: Placebo add on to valproate open label
  Placebo add on to open label valproate for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (9.5) | 41.7 (12.7) | 41.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — TimeLine Follow-Back (TLFB)
  participants
    United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Standard Drinks Per Drinking Day During the Last 4 Weeks of the Trial
Time Frame: 12 weeks
Population: One subject in the naltrexone group was considered an outlier and excluded from the analysis as it will disproportionally skew the results of small sample size, and one subject in the placebo group was lost to follow-up immediately after group allocation and before any first post allocation assessment.
Measure: Mean (Standard Deviation); unit: standard drinks/drinking day
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 8 | 8
standard drinks/drinking day | 0.6 (1.8) | 3.8 (4.2)

2. Secondary Outcome: % Subjects Abstinent
Description: Proportion of subjects abstinent during the last 4 weeks of the trial
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 9 | 9
percentage of participants | 66 | 33

ADVERSE EVENTS:
Time Frame: Adverse events reported by subjects during their participation in the study
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/9 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=9) | Placebo (N=9)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Palpitation (Cardiac disorders) | 0 (0) | 3 (3)
Nausea/ diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal cramps (Reproductive system and breast disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 2 (2)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
High early drop-out rate leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No